CLINICAL TRIAL: NCT05897658
Title: Pilot Study: Levetiracetam Prophylaxis Randomized Controlled Trial in Brain Tumor Resection
Brief Title: Levetiracetam Prophylaxis in Brain Tumor Resection Pilot
Acronym: LeviTaTe Pilot
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14147
Record Dates: First submitted 2023-04-04; First posted 2023-06-09 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Seizures; Brain Tumor
MeSH Terms: conditions — Seizures; Brain Neoplasms | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seizure Prophylaxis (Levetiracetam) (Experimental): Levetiracetam 1 g taken orally twice a day for 7 days
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator): Placebo taken orally twice a day for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Tablets
  Arms: Seizure Prophylaxis (Levetiracetam)
Other: Placebo — Tablets
  Arms: Placebo

SUMMARY:
This study aims to evaluate feasibility of a double-blind randomized controlled trial for levetiracetam prophylaxis for prevention of seizure in the perioperative phase of brain tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years or older
* Undergoing craniotomy for a brain tumor
* Intra-axial tumor location
* Supratentorial tumor location

Exclusion Criteria:

* Documented seizure history or epilepsy diagnosis
* Currently taking an antiepileptic medication
* Unable to take levetiracetam (e.g. allergy, inability to swallow)
* Inability to obtain consent from participant or substitute decision maker prior to surgery
* Renal impairment with eGFR less than 50
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, approximately 1 year
  Feasibility outcome

SECONDARY OUTCOMES:
Fraction of eligible patients approached | Through study completion, approximately 1 year
Fraction of approached patients consent | Through study completion, approximately 1 year
Role of individual who approached patients | Through study completion, approximately 1 year
  Description of research team member first approaching and consenting patients (e.g. resident, research staff, staff surgeon, etc.)
Protocol adherence | Through study completion, approximately 1 year
  Number of participants who withdrawal from the study
Protocol adherence | Through study completion, approximately 1 year
  Drug adherence rate
Protocol adherence | Through study completion, approximately 1 year
  Follow-up completion rate
Protocol adherence | Through study completion, approximately 1 year
  Method of follow-up (e.g. telephone, clinic visit)
Adverse events | Through study completion, approximately 1 year
  Serious and related adverse events and adverse drug reactions
Unblinding events | Through study completion, approximately 1 year
  Number of events and reasoning

OTHER OUTCOMES:
New onset seizure within 7 days of surgery | 7 days post-surgery, reviewed at follow-up between post-operative day 8 and 14
Incidence of infection during Study Drug administration | Follow-up between post-operative day 8 and 14
Incidence of psychiatric symptoms during Study Drug Administration | Follow-up between post-operative day 8 and 14
Length of hospital stay in days | Hospital discharge
Incidence of administration of any antiepileptic drugs | Follow-up between post-operative day 8 and 14
Incidence of administration of any benzodiazepines | Follow-up between post-operative day 8 and 14

IPD SHARING:
Plan to Share IPD: No